CLINICAL TRIAL: NCT02806232
Title: Open-label, Dose-finding, 2-parts, Efficacy Phase II Study With Three Formulations (Racemate Raziquantel Commercial Oral Tablets, New Oral Disintegrating Tablets of Racemate Praziquantel and L-praziquantel) in Schistosomiasis (S. Mansoni) Infected Children Aged 2-6 Years (Part 1), Followed by an Assessment of Efficacy and Safety With the Selected Formulation and Dosage in S. Mansoni Infected Infants Aged 3-24 Months (Part 2)
Brief Title: An Open Label Dose Finding Safety and Efficacy in Children and Infants Infected With Schistosomiasis (S.Mansoni)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200661-0005
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Schistosomiasis
Keywords: Praziquantel ODT formulation; Biltricide
MeSH Terms: conditions — Schistosomiasis | interventions — Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Part 1, Cohort 1: Biltricide (racemate praziquantel) 20 mg/kg (Experimental): Participants received Biltricide (600 mg tablet) administered orally at a dose of 20 milligram per kilogram (mg/kg), three times a day on treatment Day 1.
  Interventions: Drug: Biltricide (racemate praziquantel) oral tablets
- Part 1, Cohort 2: Biltricide (racemate praziquantel) 40 mg/kg (Experimental): Participants received Biltricide (600 mg tablet) administered orally at a dose of 40 mg/kg as a single dose on treatment Day 1.
  Interventions: Drug: Biltricide (racemate praziquantel) oral tablets
- Part 1, Cohort 3: Racemate Praziquantel 40 mg/kg (Experimental): Participants received Racemate Praziquantel oral dispersible tablet (ODT) (150 mg) administered orally at a dose of 40 mg/kg as a single dose on treatment Day 1.
  Interventions: Drug: Racemate Praziquantel ODT
- Part 1, Cohort 4: Racemate Praziquantel 60 mg/kg (Experimental): Participants received Racemate Praziquantel ODT (150 mg) administered orally at a dose of 60 mg/kg as a single dose on treatment Day 1.
  Interventions: Drug: Racemate Praziquantel ODT
- Part 1, Cohort 5: Levo Praziquantel 30 mg/kg (Experimental): Participants received Levo Praziquantel ODT (150 mg tablet) administered orally at a dose of 30 mg/kg as a single dose on treatment Day 1.
  Interventions: Drug: Levo Praziquantel ODT
- Part 1, Cohort 6: Levo Praziquantel 45 mg/kg (Experimental): Participants received Levo Praziquantel ODT (150 mg tablet) administered orally at a dose of 45 mg/kg as a single dose on treatment Day 1.
  Interventions: Drug: Levo Praziquantel ODT
- Part 1, Cohort 7: Levo Praziquantel 60 mg/kg (Experimental): Participants received Levo Praziquantel ODT (150 mg tablet) administered orally at a dose of 60 mg/kg as a single dose on treatment Day 1.
  Interventions: Drug: Levo Praziquantel ODT
- Part 2, Cohort 8: Levo Praziquantel 50 mg/kg (Experimental): Participants aged 13-24 months months received Levo Praziquantel ODT (150 mg) administered orally at a dose of 50 mg/kg as a single dose on treatment day 1.
  Interventions: Drug: Levo Praziquantel ODT
- Part 2, Cohort 9: Levo Praziquantel 50 mg/kg (Experimental): Participants aged 3 to 12 months received Levo Praziquantel ODT (150 mg) administered orally at a dose of 50 mg/kg as a single dose on treatment day 1.
  Interventions: Drug: Levo Praziquantel ODT

INTERVENTIONS:
Drug: Biltricide (racemate praziquantel) oral tablets — Biltricide (600 mg tablet) was administered to participants at a dose of 20 mg/kg in Part 1, Cohort 1 and at a dose of 40mg/kg in Part 1, Cohort 2.
  Arms: Part 1, Cohort 1: Biltricide (racemate praziquantel) 20 mg/kg; Part 1, Cohort 2: Biltricide (racemate praziquantel) 40 mg/kg
Drug: Racemate Praziquantel ODT — Racemate Praziquantel (PZQ) (150) mg was administered at a dose of 40 mg/kg in Part 1, Cohort 3 and at a dose of 60 mg/kg in Part 1, Cohort 4.
  Arms: Part 1, Cohort 3: Racemate Praziquantel 40 mg/kg; Part 1, Cohort 4: Racemate Praziquantel 60 mg/kg
Drug: Levo Praziquantel ODT — Levo PZQ (150 mg) was administered at a dose of 30 mg/kg in Part 1 Cohort 5, 45 mg/kg Part 1 Cohort 6, 60 mg/kg Part 1 Cohort 7, 50 mg/kg Part 2 Cohort 8, and 50 mg/kg Part 2 Cohort 9.
  Arms: Part 1, Cohort 5: Levo Praziquantel 30 mg/kg; Part 1, Cohort 6: Levo Praziquantel 45 mg/kg; Part 1, Cohort 7: Levo Praziquantel 60 mg/kg; Part 2, Cohort 8: Levo Praziquantel 50 mg/kg; Part 2, Cohort 9: Levo Praziquantel 50 mg/kg

SUMMARY:
The Phase II study consisted of two parts, part 1 is open label, randomized, controlled and exploratory dose finding in children aged between 2 and 6 years infected with S. mansoni. Part 2 investigated efficacy and safety with the selected formulation and dosage in S. mansoni infected children aged between 3 months - 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children aged 2 to 6 years (Part 1) and 3 to 24 months (Part 2)
* S. mansoni positive diagnosis defined as positive egg counts in stool (greater than [>]1 egg/1 occasion) according to World Health Organization (WHO) classification : light (1-99 eggs per gram of faeces), moderate (100-399 eggs per gram of faeces) and heavy (greater than or equal to [>=]400 eggs per gram of faeces) infections
* Minimum weight of 8.0 kg in 2- to 6-year-old children and of 4.0 kg in 3- to 24-month infants

  • Parents/legal representative ability to communicate well with the Investigator, to understand the protocol requirements and restrictions, and willing their children to comply with the requirements of the entire trial, i.e.
* To be examined by a study physician at screening and 14-21 days after treatment
* To provide stool and urine samples at screening, 24 hours and 8 days after treatment, as well as 14-21 days after treatment
* To provide finger prick blood samples for Pharmacokinetics (PK) studies and blood samples for safety assessments

Exclusion Criteria:

* Treatment in the 4 weeks prior to study screening with Praziquantel (PZQ) , other anti-helminthic, antimalarial or anti-retroviral compounds or any other medication that might affect the PK of PZQ such as certain antiepileptics (e.g., carbamazepine or phenytoin), glucocorticosteroids (e.g., dexamethasone), chloroquine, rifampicin or cimetidine
* For children being breast fed, treatment of the mothers/wet nurses with PZQ in the 3 days prior to administration of Investigational medicinal product
* Previous history of adverse reactions associated with PZQ treatment
* Marked increases of the liver transaminases (alanine aminotransferase and/or aspartate aminotransferase) above 3x Upper Limit of Normal (ULN)
* History of acute or severe chronic disease including hepato-splenic schistosomiasis
* Fever defined as temperature above 38.0 degree centigrade
* Debilitating illnesses such as tuberculosis, malnutrition, etc. as well as a medical history of seizures
* Mixed S. haematobium and S. mansoni infections
* Findings in the clinical examination of schistosome-infected children participating in the study as performed by the study clinician on the treatment day, that in the opinion of the Investigator constitutes a risk or a contraindication for the participation of the subject in the study or that could interfere with the study objectives, conduct or evaluation
* Unlikelihood to comply with the protocol requirements, instructions and trial-related restrictions, e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the trial

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 444 (Actual)
Dates: Start 2016-06-12 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please Contact the Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 2, Cohort 8: Levo Praziquantel 50 mg/kg: Participants aged 13-24 months received Levo Praziquantel ODT (150 mg) administered orally at a dose of 50 mg/kg as a single dose on treatment day 1.
Period: Overall Study
Arm/Group | Part 1, Cohort 1: Biltricide (Racemate Praziquantel) 20 mg/kg | Part 1, Cohort 2: Biltricide (Racemate Praziquantel) 40 mg/kg | Part 1, Cohort 3: Racemate Praziquantel 40 mg/kg | Part 1, Cohort 4: Racemate Praziquantel 60 mg/kg | Part 1, Cohort 5: Levo Praziquantel 30 mg/kg | Part 1, Cohort 6: Levo Praziquantel 45 mg/kg | Part 1, Cohort 7: Levo Praziquantel 60 mg/kg | Part 2, Cohort 8: Levo Praziquantel 50 mg/kg | Part 2, Cohort 9: Levo Praziquantel 50 mg/kg
Started | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 20 | 4
Completed | 59 | 56 | 59 | 60 | 58 | 58 | 60 | 20 | 4
Not Completed | 1 | 4 | 1 | 0 | 2 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were exposed to investigative medicinal product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, Cohort 1: Biltricide (Racemate Praziquantel) 20 mg/kg | Part 1, Cohort 2: Biltricide (Racemate Praziquantel) 40 mg/kg | Part 1, Cohort 3: Racemate Praziquantel 40 mg/kg | Part 1, Cohort 4: Racemate Praziquantel 60 mg/kg | Part 1, Cohort 5: Levo Praziquantel 30 mg/kg | Part 1, Cohort 6: Levo Praziquantel 45 mg/kg | Part 1, Cohort 7: Levo Praziquantel 60 mg/kg | Part 2, Cohort 8: Levo Praziquantel 50 mg/kg | Part 2, Cohort 9: Levo Praziquantel 50 mg/kg | Total
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 20 | 4 | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.1 (1.3) | 4.3 (1.3) | 4.4 (1.2) | 4.2 (1.2) | 4.2 (1.2) | 4.3 (1.1) | 4.4 (1.3) | 1.7 (0.3) | 0.6 (0.2) | 4.1 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 32 | 35 | 23 | 32 | 25 | 7 | 1 | 205
  Male | 38 | 32 | 28 | 25 | 37 | 28 | 35 | 13 | 3 | 239
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 20 | 4 | 444
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Cure Determined by Kato-Katz Method
Description: Clinical cure was defined as zero egg counts at 14-21 days post treatment as determined by the Kato-Katz method. Number of participants with clinical cure were reported.
Time Frame: 14-21 days post treatment
Population: Modified intention-to-treat (mITT) analysis set included all participants who had a baseline measurement for the efficacy variable and did not use anti-malaria treatment after study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort 1: Biltricide (Racemate Praziquantel) 20 mg/kg | Part 1, Cohort 2: Biltricide (Racemate Praziquantel) 40 mg/kg | Part 1, Cohort 3: Racemate Praziquantel 40 mg/kg | Part 1, Cohort 4: Racemate Praziquantel 60 mg/kg | Part 1, Cohort 5: Levo Praziquantel 30 mg/kg | Part 1, Cohort 6: Levo Praziquantel 45 mg/kg | Part 1, Cohort 7: Levo Praziquantel 60 mg/kg | Part 2, Cohort 8: Levo Praziquantel 50 mg/kg | Part 2, Cohort 9: Levo Praziquantel 50 mg/kg
Number analyzed (Participants) | 57 | 58 | 58 | 58 | 56 | 57 | 58 | 15 | 4
Participants | 51 | 43 | 47 | 46 | 44 | 49 | 52 | 14 | 4

2. Secondary Outcome: Egg Reduction Rate (Percent)
Description: Percent reduction in egg count was calculated as geometric mean egg count at post-treatment minus geometric mean egg count at baseline (before treatment) divided by geometric mean egg count at baseline.
Time Frame: Baseline, 14-21 days post treatment
Population: mITT analysis set included all participants who had a baseline measurement for the efficacy variable and did not use anti-malaria treatment after study treatment.
Measure: Geometric Mean (95% Confidence Interval); unit: percent reduction in egg count
Arm/Group | Part 1, Cohort 1: Biltricide (Racemate Praziquantel) 20 mg/kg | Part 1, Cohort 2: Biltricide (Racemate Praziquantel) 40 mg/kg | Part 1, Cohort 3: Racemate Praziquantel 40 mg/kg | Part 1, Cohort 4: Racemate Praziquantel 60 mg/kg | Part 1, Cohort 5: Levo Praziquantel 30 mg/kg | Part 1, Cohort 6: Levo Praziquantel 45 mg/kg | Part 1, Cohort 7: Levo Praziquantel 60 mg/kg | Part 2, Cohort 8: Levo Praziquantel 50 mg/kg | Part 2, Cohort 9: Levo Praziquantel 50 mg/kg
Number analyzed (Participants) | 57 | 58 | 58 | 58 | 56 | 57 | 58 | 15 | 4
percent reduction in egg count | 94.6 [89.8 to 99.4] | 83.3 [74.7 to 91.9] | 88.6 [81.8 to 95.4] | 88.6 [82.2 to 94.9] | 88.3 [81.3 to 95.3] | 92.3 [86.4 to 98.1] | 94.1 [88.6 to 99.6] | 97.7 [92.9 to 100.0] | 100.0 [100.0 to 100.0]

3. Secondary Outcome: Number of Participants With Clinical Cure Determined by Point-of-Care Circulating Cathodic Antigen (POC-CCA) Test
Description: Clinical Cure defined as no parasite eggs in the stools as assessed by the commercially available POC-CCA assay for S. mansoni. Number of participants with clinical cure were reported.
Time Frame: Day 2, Day 8 and 14-21 days post treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort 1: Biltricide (Racemate Praziquantel) 20 mg/kg | Part 1, Cohort 2: Biltricide (Racemate Praziquantel) 40 mg/kg | Part 1, Cohort 3: Racemate Praziquantel 40 mg/kg | Part 1, Cohort 4: Racemate Praziquantel 60 mg/kg | Part 1, Cohort 5: Levo Praziquantel 30 mg/kg | Part 1, Cohort 6: Levo Praziquantel 45 mg/kg | Part 1, Cohort 7: Levo Praziquantel 60 mg/kg | Part 2, Cohort 8: Levo Praziquantel 50 mg/kg | Part 2, Cohort 9: Levo Praziquantel 50 mg/kg
Number analyzed (Participants) | 57 | 58 | 58 | 58 | 56 | 57 | 58 | 15 | 4
Participants
  Day 2 | 8 | 3 | 3 | 8 | 4 | 6 | 11 | 5 | 0
  Day 8 | 28 | 16 | 19 | 18 | 16 | 28 | 38 | 8 | 0
  14-21 days post treatment | 33 | 21 | 24 | 32 | 24 | 35 | 42 | 10 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 21
Arm/Group | Part 1, Cohort 1: Biltricide (Racemate Praziquantel) 20 mg/kg | Part 1, Cohort 2: Biltricide (Racemate Praziquantel) 40 mg/kg | Part 1, Cohort 3: Racemate Praziquantel 40 mg/kg | Part 1, Cohort 4: Racemate Praziquantel 60 mg/kg | Part 1, Cohort 5: Levo Praziquantel 30 mg/kg | Part 1, Cohort 6: Levo Praziquantel 45 mg/kg | Part 1, Cohort 7: Levo Praziquantel 60 mg/kg | Part 2, Cohort 8: Levo Praziquantel 50 mg/kg | Part 2, Cohort 9: Levo Praziquantel 50 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/60 | 0/60 | 0/60 | 0/60 | 0/60 | 0/20 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/60 | 1/60 | 0/60 | 0/60 | 0/60 | 0/60 | 0/20 | 0/4
Other Adverse Events (participants affected / at risk) | 25/60 | 30/60 | 29/60 | 31/60 | 28/60 | 33/60 | 37/60 | 10/20 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, Cohort 1: Biltricide (Racemate Praziquantel) 20 mg/kg (N=60) | Part 1, Cohort 2: Biltricide (Racemate Praziquantel) 40 mg/kg (N=60) | Part 1, Cohort 3: Racemate Praziquantel 40 mg/kg (N=60) | Part 1, Cohort 4: Racemate Praziquantel 60 mg/kg (N=60) | Part 1, Cohort 5: Levo Praziquantel 30 mg/kg (N=60) | Part 1, Cohort 6: Levo Praziquantel 45 mg/kg (N=60) | Part 1, Cohort 7: Levo Praziquantel 60 mg/kg (N=60) | Part 2, Cohort 8: Levo Praziquantel 50 mg/kg (N=20) | Part 2, Cohort 9: Levo Praziquantel 50 mg/kg (N=4)
Transaminases increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, Cohort 1: Biltricide (Racemate Praziquantel) 20 mg/kg (N=60) | Part 1, Cohort 2: Biltricide (Racemate Praziquantel) 40 mg/kg (N=60) | Part 1, Cohort 3: Racemate Praziquantel 40 mg/kg (N=60) | Part 1, Cohort 4: Racemate Praziquantel 60 mg/kg (N=60) | Part 1, Cohort 5: Levo Praziquantel 30 mg/kg (N=60) | Part 1, Cohort 6: Levo Praziquantel 45 mg/kg (N=60) | Part 1, Cohort 7: Levo Praziquantel 60 mg/kg (N=60) | Part 2, Cohort 8: Levo Praziquantel 50 mg/kg (N=20) | Part 2, Cohort 9: Levo Praziquantel 50 mg/kg (N=4)
Anaemia (Blood and lymphatic system disorders) | 15 | 25 | 23 | 22 | 18 | 22 | 29 | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 3 | 3 | 5 | 4 | 0 | 6 | 1 | 0
Bronchitis (Infections and infestations) | 9 | 7 | 3 | 5 | 4 | 3 | 8 | 2 | 0
Malaria (Infections and infestations) | 5 | 3 | 5 | 1 | 4 | 4 | 2 | 5 | 1
C-reactive protein increased (Investigations) | 7 | 4 | 10 | 8 | 7 | 14 | 6 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT02806232/SAP_000.pdf
  • Study Protocol (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT02806232/Prot_001.pdf